CLINICAL TRIAL: NCT03032588
Title: A First in Human Double-blind, Randomized Study to Assess the Safety, Tolerability and Immunogenicity of a Single Dose of a Trivalent Inactivated Poliovirus Vaccine Based on Sabin Strains (sIPV) Given Intramuscularly in Healthy Adults
Brief Title: A First in Human Study to Assess the Safety, Tolerability and Immunogenicity of a Single Dose of a Trivalent Inactivated Poliovirus Vaccine Based on Sabin Strains (sIPV) Given Intramuscularly in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108290; 2016-002775-99 (EudraCT Number); GV000051POL1001 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: sIPV (Experimental): Participants will receive single intramuscular injection of the trivalent inactivated poliovirus vaccine based on Sabin strains produced on PER.C6 cells (sIPV) on Day 1.
  Interventions: Biological: sIPV
- Group 2: cIPV (Active Comparator): Participants will receive single intramuscular injection of the currently used trivalent inactivated poliovirus vaccine IMOVAX POLIO, based on the conventional Salk poliovirus strains produced on Vero cells (cIPV) on Day 1.
  Interventions: Biological: cIPV

INTERVENTIONS:
Biological: sIPV — Participants will receive single dose (0.5 milliliter [mL]) of sIPV as a suspension for intramuscular injection on Day 1.
  Other Names: JNJ-64152348
  Arms: Group 1: sIPV
Biological: cIPV — Participants will receive single dose (0.5 mL) of cIPV as a suspension for intramuscular injection on Day 1.
  Other Names: IMOVAX POLIO
  Arms: Group 2: cIPV

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of a single dose of JNJ-64152348, inactivated poliovirus vaccine produced from Sabin poliovirus strains on PER.C6 cells (sIPV) in healthy adults, using conventional inactivated poliovirus vaccine produced from Salk poliovirus strains (cIPV) as reference.

ELIGIBILITY:
Inclusion Criteria:

* Declared healthy by the investigator on the basis of physical examination, medical history, vital signs and clinical laboratory tests performed at screening. If the results of the serum chemistry panel or hematology are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Heterosexual male participants must not engage in intercourse with a female partner of childbearing potential who is not using a highly effective contraceptive method
* All female participants of childbearing potential must have a negative urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and immediately prior to study vaccine administration
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Agrees not to donate blood until the Week 4 visit

Exclusion Criteria:

* Clinically significant neuro-psychiatric, cardiovascular, pulmonary, liver or renal insufficiency (estimated creatinine clearance below 60 milliliter per minute (mL/min) using the Cockcroft-Gault Equation); metabolic, gastrointestinal, urologic, or endocrine disease that is - in the opinion of the investigator - uncontrolled
* Any history of malignancy (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Previous severe allergic reaction after vaccination with polio vaccine
* Known allergies, hypersensitivity, or intolerance to one of the excipients of JNJ-64152348, inactivated poliovirus vaccine produced from Sabin poliovirus strains on PER.C6 cells (sIPV) or conventional inactivated poliovirus vaccine produced from Salk poliovirus strains (cIPV)
* Received any polio vaccine within 6 months before study inclusion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Solicited Local Adverse Events (AEs) | Up to Day 8
  Participants will be requested to record any occurrences of solicited AEs on a daily basis in a diary on the day of dosing and during the 7 days thereafter (up to Day 8). Solicited local AEs include erythema, swelling/induration and pain/tenderness. If erythema or swelling/induration is present, the diameters will be measured using the ruler supplied and the largest diameter recorded.
Number of Participants With Solicited Systemic Adverse Events (AEs) | Up to Day 8
  Participants will be requested to record any occurrences of solicited AEs on a daily basis in a diary on the day of dosing and during the 7 days thereafter (up to Day 8). Solicited systemic AEs include fatigue, headache, nausea, myalgia and fever.
Number of Participants With Unsolicited AEs | Up to Week 4
  Unsolicited adverse events will include all adverse events for which the participant is not specifically questioned in the participant diary.
Number of Participants With Serious Adverse Events (SAEs) | Up to Week 26
  An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
Poliovirus Type- and Strain-specific Neutralizing Antibody (NAb) Responses | Up to Week 4
  Polio NAb titers will be determined against the attenuated Sabin strains (Types 1, 2 and 3) as well as against the wild-type Salk strains (Type 1 [Mahoney], Type 2 [MEF-1] and Type 3 [Saukett]), in accordance with the World Health Organization (WHO) recommendations for immunogenicity assessment of inactivated poliovirus vaccine (IPV).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Center for Vaccinology (CEVAC), Ghent, Belgium

REFERENCES:
- [Derived] Leroux-Roels I, Leroux-Roels G, Shukarev G, Schuitemaker H, Cahill C, de Rooij R, Struijs M, van Zeeburg H, Jacquet JM. Safety and immunogenicity of a new Sabin inactivated poliovirus vaccine candidate produced on the PER.C6(R) cell-line: a phase 1 randomized controlled trial in adults. Hum Vaccin Immunother. 2021 May 4;17(5):1366-1373. doi: 10.1080/21645515.2020.1812315. Epub 2020 Nov 11. PMID 33175637